CLINICAL TRIAL: NCT03519360
Title: RADAR-B: A Phase 2 Multi-center Study to Evaluate the Safety and Tolerability of Using Point-of-Care-Guided Manipulation of Ultrafiltration Rate to Prevent Hemodialysis-Associated Arrhythmias
Brief Title: Reducing Arrhythmia in Dialysis by Adjusting the Rx Electrolytes/Ultrafiltration, Study B
Acronym: RADAR-B
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties with contracting and with local dialysis unit policies preclueded successful recruiting/enrollment
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Duke University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001737-; R34HL140477-01 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: End Stage Renal Disease
Keywords: arrythmia; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restricted ultrafiltration rate (UFR) (Experimental): UFR ≤10 ml/kg/hr
  Interventions: Other: UFR-restricted dialysis
- Standard of Care/ Unrestricted UFR (Experimental): UFR as needed
  Interventions: Other: UFR-unrestricted dialysis

INTERVENTIONS:
Other: UFR-restricted dialysis — UFR's are limited to a maximum of 10 mL/kg/hr for the duration of the session. In order to prevent progressive volume overload and the need for additional hemodialysis sessions to manage volume gains in this scenario, subjects will crossover weekly between the restricted and unrestricted UFR interventions.
  Arms: Restricted ultrafiltration rate (UFR)
Other: UFR-unrestricted dialysis — UFR's will be unlimited and prescribed according to the standard of care.
  Arms: Standard of Care/ Unrestricted UFR

SUMMARY:
The purpose of this study is to test the feasibility of trials that change the dialysis ultrafiltration rate (UFR) by limiting the maximum rate and to estimate the extent to which limiting the ultrafiltration rate reduces the risk of abnormal heart rhythms in people with kidney failure who are being treated with chronic hemodialysis.

DETAILED DESCRIPTION:
Within four weeks of consent, subjects will have an Implantable Loop Recorder (ILR) (Medtronic LINQ) device implanted. Subjects will be given a transmitter/charger and a Patient Care Assistant which they will be required to keep for the duration of their participation in the study. ILR tracings will be uploaded automatically and reviewed by the study team for the occurrence of clinically significant arrhythmia.

Following ILR implantation, subjects will alternate between weekly periods in which the ultrafiltration rate can be unlimited or in which the ultrafiltration rate is limited to ≤10mL/kg/hour.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis therapy for end-stage renal disease
* Age 18-85 years (subjects between 18-40 years old will be required to have at least one of the following: history of congestive failure, diabetes, coronary or peripheral vascular disease, or arrhythmia)
* >30 days since dialysis initiation
* Ability to provide informed consent
* Interdialytic weight gain necessitating an UF rate of ≥13mL/kg/hour of dialysis to achieve the target post-dialysis weight in at least half of the dialysis sessions (≥6 sessions) in the month prior to enrollment

Exclusion Criteria:

* Expected survival <6 months-to allow trial completion
* Renal transplant, transfer to home or peritoneal dialysis, or to non-study hemodialysis facility anticipated within 6 months
* Prisoners or cognitive disability preventing informed consent
* Pregnancy. A pregnancy test will be required for women of child bearing potential prior to enrollment. A pregnancy test will not be required for women past the age of child-bearing potential >55 years old, women with a history of surgical sterilization, or for women <55 years of age who have not had a menses within the past 12 months
* Skin condition, immune dysfunction, history of multiple infections or other condition which increases risk of local infection with ILR placement
* Bleeding disorder or anti-coagulation that cannot be reversed for ILR placement
* Existing pacemaker, implantable monitor or defibrillator which precludes device placement
* Chronic, persistent AF (defined as the presence of persistent AF on all available EKGs at time of recent screening)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Adherence with Proposed Interventions | 2 years
  Adherence will be assessed as the percent of sessions in which the mandated UFR is delivered.
Incidence of unscheduled hemodialysis or hospitalization for volume overload | 4 months
  The occurrence of unscheduled hemodialysis or ultrafiltration sessions needed to treat volume overload will be measured to assess the impact of the UFR intervention on the adequacy of volume removal.
Change in duration of clinically significant arrhythmia (CSA) per month | 4 months
  The total monthly duration of CSA (in minutes) will be utilized as the primary efficacy endpoint in comparing this pair of interventions (aggressive vs. conservative UF). In the event of incomplete follow-up, CSA duration will be indexed to follow-up time. CSA will be defined on the basis of arrhythmias likely to lead to sudden cardiac arrest (SCA) or serious morbidity and mortality and will include AF, asystole ≥3 seconds, bradycardia ≤40 beats per minute lasting ≥6 seconds, and sustained VT ≥130 beats per minute lasting ≥30 seconds. CSA's will be adjudicated by study electrophysiologists.

SECONDARY OUTCOMES:
Comparison of pre- and post-correction adherence | 2 years
  This measure will assess adherence to the protocol following any corrective measures made in response to surveys of dialysis staff.
Association of individual interventions with atrial fibrillation (AF) | 4 months
  This measure will assess the effect of the interventions on the duration of atrial fibrillation.
Association of individual interventions on potentially lethal arrhythmia | 4 months
  This measure will assess the effect of the interventions on the duration of potentially lethal arrhythmias defined as asystole, sustained VT, bradycardia for ≥6 seconds.
The occurrence of clinically significant arrhythmias requiring intervention | 4 months
  This measure will assess the effect of the interventions on occurrence of arrhythmia requiring clinical intervention.
All-cause mortality | 2 years
  This measure will assess the effect of the interventions on occurrence of all-cause mortality.
Cardiovascular mortality | 2 years
  This measure will assess the effect of the interventions on occurrence of cardiovascular mortality.
Hospitalization | 2 years
  This measure will assess the effect of the interventions on occurrence of hospitalizations.
Proportion of screened patients enrolled | 2 years
  The percent of screened patients enrolled will be calculated as a secondary feasibility measure to assess the size of the necessary screening pool. Reasons for non-enrollment (vis-à-vis inclusion and exclusion criteria and patient and physician preferences) will be assessed to determine the potential for protocol modification to improve recruitment.

OTHER OUTCOMES:
Identification of barriers to implementation | 2 years
  HD staff and patients will be surveyed once 3 subjects have completed 1 month of each trial and once 6 patients have completed each trial to identify barriers to implementation of the protocol.
Association of dialysis day, shift, and site with CSA | 2 years
  Exploratory analyses will assess association of dialysis day (Monday/Wednesday/Friday or Tuesday/Thursday/Saturday), shift (1st-3rd), and site with CSA.
Association of dialysis day, shift, and site with adherence | 2 years
  Exploratory analyses will assess association of dialysis day (Monday/Wednesday/Friday or Tuesday/Thursday/Saturday), shift (1st-3rd), and site with adherence.
Association of demographic and pre-randomization factors with adverse events | 2 years
  Exploratory analyses will assess age, sex, race, mean intra-dialytic weight gain, and mean UFR in month prior to randomization on the incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD, MSc, Principal Investigator — NYU Langone Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT03519360/ICF_000.pdf